CLINICAL TRIAL: NCT02530515
Title: Trial of Immune Reconstitution With Activated T-Cells in Patients With Chronic Lymphocytic Leukemia (CLL)
Brief Title: Ex Vivo-activated Autologous Lymph Node Lymphocytes in Treating Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0830; NCI-2015-01546 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0830 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2015-08-19; First posted 2015-08-21 (Estimated); Results first posted 2019-10-29 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Anemia; Cancer Fatigue; Chronic Lymphocytic Leukemia; Fever; Infectious Disorder; Lymphadenopathy; Lymphocytosis; Night Sweats; Prolymphocytic Leukemia; Recurrent Chronic Lymphocytic Leukemia; Richter Syndrome; Secondary Malignant Neoplasm; Thrombocytopenia; Weight Loss
MeSH Terms: conditions — Anemia; Leukemia, Lymphocytic, Chronic, B-Cell; Fever; Communicable Diseases; Lymphadenopathy; Lymphocytosis; Leukemia, Prolymphocytic; Neoplasms, Second Primary; Thrombocytopenia; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ex vivo autologous lymph node lymphocytes) (Experimental): Patients receive infusion of ex vivo-activated autologous lymph node lymphocytes IV over 10-30 minutes on day 0.
  Interventions: Biological: Ex Vivo-activated Autologous Lymph Node Lymphocytes; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Ex Vivo-activated Autologous Lymph Node Lymphocytes — Given IV
  Other Names: X-ACT; X-ACT Autologous Lymph Node Lymphocytes
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies the side effects of ex vivo-activated autologous lymph node lymphocytes infusion and to see how well they work in treating patients with chronic lymphocytic leukemia. Biological therapies, such as ex vivo-activated autologous lymph node lymphocytes, use substances made from living organisms that may stimulate or suppress the immune system in different ways and stop tumor cells from growing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility and safety of infusion of autologous activated T-cells (ex vivo-activated autologous lymph node lymphocytes) in patients with chronic lymphocytic leukemia.

SECONDARY OBJECTIVES:

I. To study immune reconstitution following infusion of activated T-cells in patients with chronic lymphocytic leukemia.

II. To study the incidence of infections for up to 1 year following activated T cell infusion.

III. To study the overall response rates.

OUTLINE:

Patients receive infusion of ex vivo-activated autologous lymph node lymphocytes intravenously (IV) over 10-30 minutes on day 0.

Patients who have been previously treated on study, and subsequently need additional infusions, may be retreated with previously cryopreserved expanded cells at the same or lower dose level 6-12 months after the first infusion.

After completion of study treatment, patients are followed up at 1.5 years and then every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a diagnosis of chronic lymphocytic leukemia (CLL) by immunophenotyping and flow cytometry analysis of blood or bone marrow

  * Patients must meet criteria for treatment based on the criteria proposed by National Cancer Institute (NCI)-sponsored CLL Working Group to include at least one of the following:

    * Weight loss of more than 10% over the preceding 6 months; or
    * Extreme fatigue attributable to progressive disease; or
    * Fever or night sweats without evidence of infection; or
    * Worsening anemia (Rai stage Ill) or thrombocytopenia (Rai stage IV); or
    * Massive lymphadenopathy (> 10 cm) or rapidly progressive lymphocytosis (lymphocyte doubling time < 6 months); or
    * Prolymphocytic or Richter's transformation; or
  * Patients with CLL who have received at least one prior line of therapy; or
  * Patients with CLL who have frequent infections and/or recurrent secondary cancers
* No active central nervous system (CNS) disease
* All patients must have a Karnofsky performance score > 60%
* Calculated creatinine clearance (by Cockcroft-Gault) of > 50 ml/min
* Patients must not have untreated or uncontrolled life-threatening infection
* Patients must sign informed consent

Exclusion Criteria:

* Receipt of glucocorticoids (with the exception of inhaled glucocorticoid steroids for the use of allergic rhinitis or pulmonary disease) within 2 weeks of registration
* Autoimmune disease related to CLL, e.g., idiopathic thrombocytopenic purpura (ITP) or autoimmune hemolytic anemia, is permitted if not requiring active treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-12-18 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chitra Hosing, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients who qualify for lymphodepleting chemotherapy and who do not have 17p deletion are randomized to Arm A or Arm B. Those patients who do not qualify by those criteria are assigned to Arm C.
Groups:
- Arm A: Receive lymphodepletion chemotherapy followed by activated T-cell infusion
- Arm B: Receive lymphodepletion chemotherapy followed by activated T-cell infusion followed by low dose lenalidomide PO once ANC is>1.5x109/L
- Arm C: Patients who cannot receive lymphodepleting chemotherapy (as determined by the treating physician) or those with 17p deletion
Period: Overall Study
Arm/Group | Arm A | Arm B | Arm C
Started | 0 | 0 | 8
Completed | 0 | 0 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients were enrolled in Arm C at the physician's discretion and there is no analysis to compare between the lenalidomide Arm A vs the non-lenalidomide Arm B
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Arm C | Total
Number analyzed (Participants) | 0 | 0 | 8 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 1 | 1
  >=65 years | 0 | 0 | 7 | 7
Age, Continuous [Median (Full Range); unit: years] |  |  | 74.5 [64 to 84] | 74.5 [64 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 4 | 4
  Male | 0 | 0 | 4 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 7 | 7
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 7 | 7
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success and Feasibility of Autologous Activated T-cells Infusion, Determined by Number of Participants That Achieved Target-Activated T-cell Dose Without DLT.
Description: Success will be defined as achievement of a target activated T-cell dose of 1x108 +/-20% without DLT and the lack of dose limiting toxicity (DLT). DLT for this trial is defined as any Grade 4 or higher non-hematologic toxicity or grade 3 or 4 allergy/immunology toxicity, allergic reaction or urticaria grade 3 or higher by +90 days after T cell infusion, Grade 2 or greater autoimmune phenomena, or Grade 4 or higher hematologic toxicity (with the exception of any preexisting AE due to prior treatment or due to disease) deemed related to T cells and occurring by day +90 after T cell infusion. Feasibility is defined as achievement of the target T-cell dose (1x108 +/-20% ) without DLT in >50% of patients enrolled.
Time Frame: Enrollment up to day 100 post T cell infusion for each arm.
Population: Patients with CLL.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 0 | 0 | 8
Participants
  Sucessful Target T-cell Dose |  |  | 7
  Feasibility |  |  | 7

2. Secondary Outcome: Immune Reconstitution
Description: To study immune reconstitution following infusion of activated T-cells in patients with chronic lymphocytic leukemia
Time Frame: Up to 1 year
Population: Data was not collected due to low accrual
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Overall Response Rates
Description: The overall response rates between the lenalidomide and non-lenalidomide arms. For response to treatment, it was measured by International Workshop on CLL (iwCLL), criteria 2008 guidelines.
Time Frame: Up to 1 year
Population: Data was not collected due to low accrual
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Incidence of Infections
Description: To study the incidence of infections for up to 1 year following activated T cell infusion
Time Frame: Up to 1 year
Population: Data was not collected due to low accrual
Arm/Group | Arm A | Arm B | Arm C
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 100 Days post T cell infusion.
Description: Patients who qualify for lymphodepleting chemotherapy and who do not have 17p deletion are randomized to Arm A or Arm B. Those patients who do not qualify by those criteria are assigned to Arm C.
Arm/Group | Arm A | Arm B | Arm C
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/8
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=0) | Arm B (N=0) | Arm C (N=8)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 (4)
Hypertension (Cardiac disorders) | 0 | 0 | 1 (1)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 (2)
Platelet Count Decreased (Investigations) | 0 | 0 | 2 (2)
Eye Infection (Infections and infestations) | 0 | 0 | 1 (1)
Mucositis (Gastrointestinal disorders) | 0 | 0 | 1 (1)
Nail Infection (Infections and infestations) | 0 | 0 | 1 (1)
Sinusitis (Infections and infestations) | 0 | 0 | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 3 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 (1)
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1)
Edema limbs (General disorders) | 0 | 0 | 1 (1)
Fatigue (General disorders) | 0 | 0 | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 (1)
Skin Other (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT02530515/Prot_SAP_000.pdf